CLINICAL TRIAL: NCT01511250
Title: A Double-Blind, Randomized, Placebo-Controlled, Age Descending and Expansion Phase 2 Study to Investigate the Safety and Immunogenicity of a Tetravalent Chimeric Dengue Vaccine in Healthy Volunteers Between the Ages of 1.5 - 45 Years
Brief Title: Study to Investigate the Safety and Immunogenicity of a Tetravalent Chimeric Dengue Vaccine in Healthy Volunteers Between the Ages of 1.5 - 45 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INV-DEN-203; 2022-003455-33 (EudraCT Number)
Record Dates: First submitted 2011-11-16; First posted 2012-01-18 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: Normal healthy adults and children; Safety and tolerability; Active vaccine; Placebo; Dengue virus vaccine; Immune response

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part I: TDV 21 to 45 Years (yrs) (Experimental): TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose). TDV comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4 containing 2*10^4 plaque forming units (PFU), 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU respectively, total virus per dose: 4.7*10^5 PFU.
  Interventions: Biological: TDV
- Part I: Placebo 21 to 45 yrs (Placebo Comparator): TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose).
  Interventions: Biological: Placebo
- Part I: TDV 12 to 20 yrs (Experimental): TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose). TDV comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4 containing 2*10^4 PFU, 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU respectively, total virus per dose: 4.7*10^5 PFU.
  Interventions: Biological: TDV
- Part I: Placebo 12 to 20 yrs (Placebo Comparator): TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose).
  Interventions: Biological: Placebo
- Part I: TDV 6 to 11 yrs (Experimental): TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose). TDV comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4 containing 2*10^4 PFU, 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU respectively, total virus per dose: 4.7*10^5 PFU.
  Interventions: Biological: TDV
- Part I: Placebo 6 to 11 yrs (Placebo Comparator): TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose).
  Interventions: Biological: Placebo
- Part I: TDV 1.5 to 5 yrs (Experimental): TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose). TDV comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4 containing 2*10^4 PFU, 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU respectively, total virus per dose: 4.7*10^5 PFU.
  Interventions: Biological: TDV
- Part I: Placebo 1.5 to 5 yrs (Placebo Comparator): TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose).
  Interventions: Biological: Placebo
- Part II: TDV 1.5 to 11 yrs (Experimental): TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose). TDV comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4 containing 2*10^4 PFU, 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU respectively, total virus per dose: 4.7*10^5 PFU.
  Interventions: Biological: TDV
- Part II: Placebo 1.5 to 11 yrs (Placebo Comparator): TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TDV — TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose). TDV comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4 containing 2*10^4 PFU, 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU respectively, total virus per dose: 4.7*10^5 PFU.
  Arms: Part I: TDV 1.5 to 5 yrs; Part I: TDV 12 to 20 yrs; Part I: TDV 21 to 45 Years (yrs); Part I: TDV 6 to 11 yrs; Part II: TDV 1.5 to 11 yrs
Biological: Placebo — TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose).
  Arms: Part I: Placebo 1.5 to 5 yrs; Part I: Placebo 12 to 20 yrs; Part I: Placebo 21 to 45 yrs; Part I: Placebo 6 to 11 yrs; Part II: Placebo 1.5 to 11 yrs

SUMMARY:
The purpose of this study is to assess the safety of Takeda's tetravalent dengue vaccine (TDV) (previously DENVax) administered subcutaneously in healthy adults and children. In addition the antibody response to the four dengue virus serotypes will be evaluated.

DETAILED DESCRIPTION:
The vaccine tested in this study was tetravalent dengue vaccine (TDV). TDV was tested to assess safety and immunogenicity in healthy adults and children living in dengue endemic countries.

The study enrolled 360 healthy participants. The study was conducted in 2 parts, Part 1 - age descending and and Part 2 - expansion - ages 1.5-11 years. Participants were allocated to one of the four age cohorts in Part 1 (21 to 45 years, 12 to 20 years, 6 to 11 years, and 1.5 to 5 years) and expansion age cohort 1.5-11 years in Part 2. Participants were randomized in 2:1 ratio and in 3: 1 ratio in Part 1 and 2 respectively to receive:

* TDV 0.5 mL SC injection
* Placebo (inactive solution) - this is a solution that looks like the study drug but has no active ingredient

This multi-center trial was conducted worldwide. The overall time to participate in this study was up to 37 months (including screening period). Participants made multiple visits to the clinic including a final visit at Day 1080.

ELIGIBILITY:
Inclusion Criteria:

* In good health as determined by medical history, physical examination including height and weight
* Normal safety laboratory values at screening
* Negative for human immunodeficiency virus-1 (HIV-1) antibodies, Hepatitis C antibodies & Hepatitis B surface antigen
* Females negative by urine pregnancy test at screening and immediately prior to injection, and were willing to use reliable means of contraception
* Weight: Within 1.3 times of the upper limit of local normal age-adjusted body mass index (BMI)

Exclusion Criteria:

* For participants ≥12 years, clinically significant electrocardiogram (ECG) findings
* History of significant dermatologic (skin) disease within last 6 months
* History of diabetes mellitus
* History of thymic pathology, thymectomy, myasthenia or any immunodeficiency
* History of recurring headaches or migraines
* Hypersensitivity to any vaccine
* For participants ≥12 years, positive urine screen for cocaine, amphetamines, opiates, or cannabinoids
* History of alcohol abuse
* Pregnant or lactating female

Ages: 18 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2011-11-16 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (8):
- Program For The Study and Control of Tropical Diseases, Medellín, Colombia
- Puerto Rico (3):
  - Ponce School of Medicine, CAIMED Center, Ponce
  - University of Puerto Rico School of Medicine, San Juan
  - Latin Clinical Trial Center, San Juan
- Singapore (2):
  - National University Hospital, Singapore
  - Changi General Hospital, Singapore
- Thailand (2):
  - Faculty of Tropical Medicine, Mahidol University, Bangkok, Bangkok
  - Phramongkutklao Hospital, Bangkok, Bangkok

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800
- [Derived] Nascimento EJM, Norwood B, Kpamegan E, Parker A, Fernandes J, Perez-Guzman E, Tricou V, Braun R, Sharma M, Dean HJ. Antibodies Produced in Response to a Live-Attenuated Dengue Vaccine Are Functional in Activating the Complement System. J Infect Dis. 2023 May 29;227(11):1282-1292. doi: 10.1093/infdis/jiac476. PMID 36461942
- [Derived] Tsuji I, Dominguez D, Egan MA, Dean HJ. Development of a Novel Assay to Assess the Avidity of Dengue Virus-Specific Antibodies Elicited in Response to a Tetravalent Dengue Vaccine. J Infect Dis. 2022 May 4;225(9):1533-1544. doi: 10.1093/infdis/jiab064. PMID 33534885
- [Derived] Sirivichayakul C, Barranco-Santana EA, Rivera IE, Kilbury J, Raanan M, Borkowski A, Papadimitriou A, Wallace D. Long-term Safety and Immunogenicity of a Tetravalent Dengue Vaccine Candidate in Children and Adults: A Randomized, Placebo-Controlled, Phase 2 Study. J Infect Dis. 2022 May 4;225(9):1513-1520. doi: 10.1093/infdis/jiaa406. PMID 32658250
- [Derived] Sharma M, Glasner DR, Watkins H, Puerta-Guardo H, Kassa Y, Egan MA, Dean H, Harris E. Magnitude and Functionality of the NS1-Specific Antibody Response Elicited by a Live-Attenuated Tetravalent Dengue Vaccine Candidate. J Infect Dis. 2020 Mar 2;221(6):867-877. doi: 10.1093/infdis/jiz081. PMID 30783676
- [Derived] Rupp R, Luckasen GJ, Kirstein JL, Osorio JE, Santangelo JD, Raanan M, Smith MK, Wallace D, Gordon GS, Stinchcomb DT. Safety and immunogenicity of different doses and schedules of a live attenuated tetravalent dengue vaccine (TDV) in healthy adults: A Phase 1b randomized study. Vaccine. 2015 Nov 17;33(46):6351-9. doi: 10.1016/j.vaccine.2015.09.008. Epub 2015 Sep 15. PMID 26384447
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b60244db2bf003ab4974e?idFilter=%5B%22DEN-313%22%2C%22INV-DEN-203%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in Puerto Rico, Colombia, Singapore and Thailand from 16 November 2011 to 15 April 2016.
Pre-assignment Details: Healthy participants were enrolled in the 2-part study to receive 0.5 mL tetravalent dengue vaccine (TDV) or placebo in 1 of 4 groups for Part I: 21-45 years, 12-20 years, 6-11 years, 1.5-5 years, and in 1 group for Part II: 1.5-11 years. Part II started after all subjects in Part 1 were enrolled.
Groups:
- Part I: TDV 21 to 45 Years: TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose) in participants aged 21 to 45 years. TDV comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4 containing 2*10^4 plaque forming units (PFU), 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU respectively, total virus per dose: 4.7*10^5 PFU.
- Part I: Placebo 21 to 45 Years: TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose) in participants aged 21 to 45 years.
- Part I: TDV 12 to 20 Years: TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose) in participants aged 12 to 20 years. TDV comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4 containing 2*10^4 PFU, 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU respectively, total virus per dose: 4.7*10^5 PFU.
- Part I: Placebo 12 to 20 Years: TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose) in participants aged 12 to 20 years.
- Part I: TDV 6 to 11 Years: TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose) in participants aged 6 to 11 years. TDV comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4 containing 2*10^4 PFU, 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU respectively, total virus per dose: 4.7*10^5 PFU.
- Part I: Placebo 6 to 11 Years: TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose) in participants aged 6 to 11 years.
- Part I: TDV 1.5 to 5 Years: TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose) in participants aged 1.5 to 5 years. TDV comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4 containing 2*10^4 PFU, 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU respectively, total virus per dose: 4.7*10^5 PFU.
- Part I: Placebo 1.5 to 5 Years; Part II: Placebo 1.5 to 11 Years: TDV placebo-matching 0.5 mL injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose) in participants aged 1.5 to 5 years.
- Part II: TDV 1.5 to 11 Years: TDV 0.5 mL, injection, subcutaneously, once on Day 0 (first dose) and Day 90 (second dose) in participants aged 1.5 to 11 years. TDV comprised of 4 recombinant, live attenuated dengue virus strains: TDV-1, TDV-2, TDV-3 and TDV-4 containing 2*10^4 PFU, 5*10^4 PFU, 1*10^5 PFU, and 3*10^5 PFU respectively, total virus per dose: 4.7*10^5 PFU.
Period: Overall Study
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Started | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53
Completed | 15 | 9 | 18 | 11 | 21 | 17 | 21 | 9 | 145 | 48
Not Completed | 9 | 5 | 4 | 3 | 0 | 0 | 2 | 4 | 14 | 5
Not completed — Withdrawal of Consent | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Sponsor/Investigator Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 3 | 3 | 3 | 0 | 0 | 2 | 3 | 13 | 5
Not completed — Protocol Violation | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received at least one dose of study vaccine or placebo and for whom valid pre-dosing and at least one valid post-dosing blood sample have been received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years | Total
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53 | 360
Age, Continuous [Mean (Full Range); unit: years] | 29.2 [21.0 to 45.0] | 30.1 [21.0 to 40.0] | 15.5 [12.0 to 19.0] | 16.8 [12.0 to 20.0] | 8.4 [6.0 to 11.0] | 7.8 [6.0 to 11.0] | 3.3 [1.5 to 5.0] | 3.5 [2.3 to 5.0] | 6.6 [1.6 to 11.0] | 6.8 [2.1 to 11.0] | 9.8 [1.5 to 45.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 12 | 7 | 6 | 8 | 7 | 7 | 88 | 19 | 172
  Male | 14 | 6 | 10 | 7 | 15 | 9 | 16 | 6 | 71 | 34 | 188
Race [Number; unit: participants]
  Asian | 3 | 3 | 16 | 8 | 16 | 12 | 12 | 6 | 77 | 24 | 177
  Hispanic or Latino | 20 | 10 | 6 | 6 | 4 | 5 | 11 | 7 | 79 | 27 | 175
  White | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 5
Seropositive to any Serotype at Day 0 [Number; unit: participants] — Seropositivity is defined as a reciprocal neutralizing titer measured by a microneutralizing test 50% (MNT50) greater or equal to (≥)10.
  participants
    Seropositive to any Serotype=No | 5 | 2 | 7 | 1 | 12 | 14 | 16 | 12 | 93 | 24 | 186
    Seropositive to any Serotype=Yes | 19 | 12 | 15 | 13 | 9 | 3 | 7 | 1 | 66 | 29 | 174
Height [Mean (Full Range); unit: meters (m)] | 1.68 [1.57 to 1.82] | 1.65 [1.53 to 1.87] | 1.58 [1.38 to 1.72] | 1.60 [1.41 to 1.73] | 1.29 [1.08 to 1.52] | 1.27 [1.13 to 1.42] | 0.98 [0.83 to 1.13] | 0.99 [0.90 to 1.06] | 1.20 [0.77 to 1.62] | 1.22 [0.83 to 1.63] | 1.28 [0.77 to 1.87]
Weight [Mean (Full Range); unit: kilograms (kg)] | 81.6 [41.4 to 115.1] | 80.2 [56.3 to 120.4] | 57.0 [28.6 to 93.4] | 59.5 [48.6 to 89.9] | 31.2 [18.5 to 51.2] | 27.0 [20.3 to 37.5] | 15.1 [10.3 to 22.2] | 16.5 [13.3 to 20.8] | 25.7 [10.4 to 61.0] | 26.7 [10.6 to 53.2] | 34.3 [10.3 to 120.4]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 28.81 [14.70 to 41.30] | 29.05 [21.30 to 38.70] | 22.60 [15.00 to 33.60] | 23.09 [18.60 to 31.50] | 18.38 [12.90 to 28.80] | 16.56 [14.20 to 20.60] | 15.63 [12.50 to 19.00] | 16.95 [13.20 to 20.40] | 17.02 [12.10 to 30.10] | 17.08 [13.20 to 24.30] | 18.83 [12.10 to 41.30]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary-Recorded) Following Either Vaccination Dose by Severity
Description: Solicited local injection site reactions were collected by subject diary and graded based on the Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03 for pain [Grade 0 (no pain), 1 (mild), 2 (moderate) and 3 (severe)] and itching (pruritus) [Grade 0 (no itching), 1 (mild), 2 (moderate) and 3 (Severe]. Severity grade for redness (erythema) and swelling (edema/induration) were derived from recorded length of the longest diameter measurement using the FDA Guidance for Industry: Toxicity Grading Scale of Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trial were Grade 0 (<2.5 cm), 1 (mild: 2.5-5 cm), 2 (moderate: 5.1-10 cm) and 3 (severe: >10 cm) and Grade 4 (Potentially Life-threatening: necrosis or exfoliative dermatitis).
Time Frame: Within 14 days after either of the vaccination given on Day 0 or 90 (Day 14 for first vaccination, Day 104 for second vaccination)
Population: The safety set included all randomized participants who received at least one dose of study vaccine (or placebo). Only categories for which there was at least 1 participant are reported.
Measure: Number; unit: participants
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53
participants
  Pain, Any Severity | 7 | 0 | 14 | 3 | 9 | 0 | 7 | 2 | 56 | 6
  Pain, Grade 1 | 7 | 0 | 11 | 2 | 4 | 0 | 7 | 2 | 41 | 3
  Pain, Grade 2 | 0 | 0 | 3 | 1 | 4 | 0 | 0 | 0 | 11 | 3
  Pain, Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0
  Itching, Any Severity | 3 | 1 | 7 | 1 | 2 | 1 | 2 | 0 | 26 | 4
  Itching, Grade 1 | 3 | 1 | 7 | 1 | 1 | 1 | 2 | 0 | 19 | 3
  Itching, Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 1
  Itching, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Erythema, Any Severity | 6 | 0 | 4 | 0 | 2 | 0 | 3 | 0 | 24 | 1
  Erythema, Grade 1 | 5 | 0 | 4 | 0 | 1 | 0 | 3 | 0 | 21 | 0
  Erythema, Grade 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Erythema, Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Edema, Any Severity | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 13 | 0
  Edema, Grade 1 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 9 | 0
  Edema, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Edema, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (In Clinic Assessment) Following Either Vaccination Dose by Severity
Description: as for outcome 1
Time Frame: Within 28 days after either of the vaccination given on Day 0 or 90 (Day 28 for first vaccination, Day 118 for second vaccination)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53
participants
  Pain, Any Severity | 2 | 0 | 4 | 2 | 9 | 5 | 5 | 1 | 33 | 14
  Pain, Grade 1 | 2 | 0 | 3 | 2 | 9 | 5 | 5 | 1 | 28 | 13
  Pain, Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1
  Itching, Any Severity | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 4 | 5
  Itching, Grade 1 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 4 | 5
  Erythema, Any Severity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema, Any Severity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events (AEs) (Diary-Recorded) Following Either Vaccination Dose by Severity
Description: Solicited systemic AEs (headache, muscle pain [myalgia], joint pain [arthralgia], eye pain, sensitivity to light [photophobia], tiredness [fatigue], body rash, nausea, were recorded in the participant's-diary along with vomiting [number of times]), and body temperature). Diary-recorded severity grades were based on the Common Terminology Criteria for Adverse Events (CTCAE). Severity grades were: Mild (Grade 1): transient symptoms, discomfort noticed but was easily tolerated by the participant with no interference to normal daily activities. Moderate (Grade 2): marked symptoms, moderate interference with participant's daily activities. Severe (Grade 3): Considerable interference with participant's daily activities. The CTCAE severity grades for fever and vomiting were derived from the diary-recorded measurements of temperature level and number of episodes, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53
participants
  Fever, Any Severity | 1 | 3 | 4 | 1 | 1 | 1 | 4 | 4 | 33 | 9
  Fever, Grade 1 | 0 | 1 | 4 | 1 | 1 | 1 | 4 | 2 | 27 | 6
  Fever, Grade 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 2
  Fever, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Headache, Any Grade | 6 | 4 | 9 | 8 | 4 | 5 | 3 | 4 | 46 | 12
  Headache, Grade 1 | 3 | 1 | 4 | 5 | 3 | 3 | 3 | 3 | 30 | 6
  Headache, Grade 2 | 2 | 2 | 5 | 3 | 1 | 2 | 0 | 1 | 12 | 4
  Headache, Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Myalgia, Any Severity | 4 | 3 | 4 | 5 | 1 | 3 | 5 | 2 | 30 | 6
  Myalgia, Grade 1 | 3 | 1 | 2 | 2 | 1 | 3 | 3 | 0 | 21 | 4
  Myalgia, Grade 2 | 0 | 1 | 2 | 2 | 0 | 0 | 2 | 1 | 6 | 1
  Myalgia, Grade 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1
  Arthralgia, Any Severity | 1 | 3 | 2 | 2 | 0 | 0 | 1 | 1 | 10 | 2
  Arthralgia, Grade 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 7 | 1
  Arthralgia, Grade 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 1
  Arthralgia, Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Eye Pain, Any Severity | 3 | 3 | 1 | 3 | 0 | 0 | 2 | 1 | 14 | 3
  Eye Pain, Grade 1 | 1 | 2 | 0 | 2 | 0 | 0 | 2 | 1 | 11 | 3
  Eye Pain, Grade 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0
  Eye Pain, Grade 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Photophobia, Any Severity | 3 | 1 | 0 | 4 | 1 | 0 | 0 | 0 | 11 | 3
  Photophobia, Grade 1 | 1 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 9 | 3
  Photophobia, Grade 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
  Photophobia, Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue, Any Severity | 4 | 4 | 9 | 6 | 2 | 5 | 3 | 3 | 29 | 10
  Fatigue, Grade 1 | 2 | 2 | 7 | 2 | 1 | 2 | 1 | 2 | 19 | 6
  Fatigue, Grade 2 | 0 | 0 | 2 | 4 | 0 | 3 | 2 | 0 | 7 | 3
  Fatigue, Grade 3 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1
  Body rash, Any Severity | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 2 | 14 | 2
  Body rash, Grade 1 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 2 | 12 | 2
  Body rash, Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Body rash, Grade 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Nausea, Any Severity | 4 | 1 | 3 | 4 | 1 | 0 | 3 | 3 | 22 | 4
  Nausea, Grade 1 | 2 | 1 | 3 | 2 | 0 | 0 | 2 | 3 | 14 | 4
  Nausea, Grade 2 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 4 | 0
  Nausea, Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
  Vomiting, Any Severity | 2 | 1 | 0 | 2 | 1 | 1 | 4 | 5 | 18 | 3
  Vomiting, Grade 1 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 2 | 5 | 2
  Vomiting, Grade 2 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 11 | 1
  Vomiting, Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

4. Primary Outcome: Number of Participants With Any Solicited AE Following Either Vaccination Dose
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. Solicited local injection site reactions included pain, itching, erythema, edema and solicited systemic AEs include myalgia, arthralgia, eye pain, photophobia, fatigue, body rash, nausea, vomiting, and fever.
Time Frame: as for outcome 1
Population: The safety set included all randomized participants who received at least one dose of study vaccine (or placebo).
Measure: Number; unit: participants
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53
participants | 13 | 9 | 17 | 12 | 12 | 8 | 17 | 10 | 110 | 28

5. Primary Outcome: Number of Participants With at Least One Unsolicited AE Following Either Vaccination Dose by Severity
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. The severity of all unsolicited AEs was evaluated by the Investigator (using the Common Terminology Criteria for Adverse Events [CTCAE] v4.03) as follows. Mild (Grade 1): Transient symptoms, discomfort noticed but was easily tolerated by the participant with no interference to normal daily activities. Moderate (Grade 2): Marked symptoms, moderate interference with participant's daily activities. Severe (Grade 3): Considerable interference with participant's daily activities.
Time Frame: Unsolicited AEs were collected within 28 days of all vaccinations. Serious AEs were collected throughout the study up to Day 1080
Population: The safety set included all randomized participants who received at least one dose of study vaccine (or placebo).
Measure: Number; unit: participants
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53
participants
  At least one unsolicited AE | 13 | 7 | 14 | 8 | 12 | 11 | 17 | 12 | 101 | 37
  Unsolicited AEs by worst severity, Mild | 6 | 2 | 7 | 2 | 10 | 8 | 13 | 10 | 72 | 31
  Unsolicited AEs by worst severity, Moderate | 5 | 5 | 6 | 5 | 1 | 3 | 4 | 2 | 25 | 6
  Unsolicited AEs by worst severity, Severe | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 4 | 0

6. Primary Outcome: Seropositivity Rate to Each of the Four Dengue Serotypes at Day 120
Description: Seropositivity rate, defined as the percentage of participants seropositive, was derived from titers of dengue-neutralizing antibodies. Participants were classified by titer after Day 0 as seropositive or seronegative. Seropositive was defined as a MNT50 titre value of ≥10 for any serotype and seronegative was defined as titre value of less than (<) 10 for all 4 serotypes. Seropositivity was assessed for the four dengue serotypes: TDV-1, TDV-2, TDV-3, TDV-4.
Time Frame: 30 days after second vaccination (Day 120)
Population: FAS included all randomized participants who received at least one dose of study vaccine or placebo and for whom valid pre-dosing and at least one valid post-dosing blood sample has been received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
percentage of participants
  TDV-1 | 100.0 [84.6 to 100.0] | 92.3 [64 to 99.8] | 100.0 [84.6 to 100.0] | 85.7 [57.2 to 98.2] | 100.0 [83.9 to 100.0] | 23.5 [6.8 to 49.9] | 100.0 [84.6 to 100.0] | 0.0 [0.0 to 28.5] | 100.0 [97.7 to 100.0] | 43.4 [29.8 to 57.7]
  TDV-2 | 100.0 [84.6 to 100.0] | 84.6 [54.6 to 98.1] | 95.5 [77.2 to 99.9] | 85.7 [57.2 to 98.2] | 100.0 [83.9 to 100.0] | 23.5 [6.8 to 49.9] | 100.0 [84.6 to 100.0] | 0.0 [0.0 to 28.5] | 100.0 [97.7 to 100.0] | 35.8 [23.1 to 50.2]
  TDV-3 | 100.0 [84.6 to 100.0] | 100.0 [75.3 to 100.0] | 100.0 [84.6 to 100.0] | 85.7 [57.2 to 98.2] | 100.0 [83.9 to 100.0] | 29.4 [10.3 to 56] | 100.0 [84.6 to 100.0] | 0.0 [0.0 to 28.5] | 99.4 [96.5 to 100.0] | 35.8 [23.1 to 50.2]
  TDV-4 | 90.9 [70.8 to 98.9] | 61.5 [31.6 to 86.1] | 72.7 [49.8 to 89.3] | 71.4 [41.9 to 91.6] | 85.7 [63.7 to 97.0] | 29.4 [10.3 to 56.0] | 100.0 [84.6 to 100.0] | 0.0 [0.0 to 28.5] | 94.9 [90.1 to 97.8] | 35.8 [23.1 to 50.2]

7. Secondary Outcome: Part I: Number of Participants Positive for Vaccine Viremia for Each of Four Vaccine Strain Serotypes After the Each Vaccination
Description: Vaccine viremia was assessed for each of the four vaccine strain serotypes: TDV-1, TDV-2, TDV-3 and TDV-4 for Part-1. Vaccine viral ribonucleic acid (RNA) was detected by a quantitative reverse transcription-polymerase chain reaction (qRT-PCR) assay.
Time Frame: Days 0, 7, 14, 90, 97, and 104
Population: The FAS included all randomized participants who received at least one dose of study vaccine and for whom valid pre-dosing and at least one valid post-dosing blood sample have been received.
Measure: Number; unit: participants
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13
participants
  Day 0, TDV-1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 0, TDV-2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 0, TDV-3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 0, TDV-4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7, TDV-1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7, TDV-2 | 2 | 0 | 4 | 0 | 4 | 0 | 9 | 0
  Day 7, TDV-3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7, TDV-4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14, TDV-1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14, TDV-2 | 0 | 0 | 3 | 0 | 6 | 0 | 4 | 0
  Day 14, TDV-3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14, TDV-4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 90, TDV-1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 90, TDV-2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 90, TDV-3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 90, TDV-4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 97, TDV-1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 97, TDV-2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Day 97, TDV-3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 97, TDV-4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 104, TDV-1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 104, TDV-2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Day 104, TDV-3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 104, TDV-4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Part I: Duration of Vaccine Viremia
Time Frame: Days 0, 7, 14, 90, 97, and 104
Population: Due to the very low prevalence of vaccine viremia, there was insufficient data for the estimation of average titer duration of viral RNA within study groups.
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Part I: Titers of Vaccine Viremia
Time Frame: Days 0, 7, 14, 90, 97, and 104
Population: as for outcome 8
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Seropositivity Rate to Each of the Four Dengue Serotypes
Description: Seropositivity rate, defined as the percentage of participants seropositive, was derived from titers of dengue-neutralizing antibodies. Participants were classified by titer after Day 0 as seropositive or seronegative. Seropositive was defined as a MNT50 titre value of ≥10 and seronegative was defined as titre value of less than (<) 10. Seropositivity was assessed for the four dengue serotypes: TDV-1, TDV-2, TDV-3, TDV-4.
Time Frame: Day 28 and Day 90 (Parts 1 and 2) and Days 180, 360, 720 and 1080 in Part 1
Population: FAS included all randomized participants who received at least one dose of study vaccine or placebo and for whom valid pre-dosing and at least one valid post-dosing blood sample have been received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53
percentage of participants
  Day 28, TDV-1: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-1 | 100.0 [85.8 to 100.0] | 92.3 [64.0 to 99.8] | 86.4 [65.1 to 97.1] | 85.7 [57.2 to 98.2] | 100.0 [83.9 to 100.0] | 23.5 [6.8 to 49.9] | 100.0 [85.2 to 100.0] | 7.7 [0.2 to 36.0] | 100.0 [97.7 to 100.0] | 41.5 [28.1 to 55.9]
  Day 28, TDV-2: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-2 | 100.0 [85.8 to 100.0] | 92.3 [64.0 to 99.8] | 86.4 [65.1 to 97.1] | 85.7 [57.2 to 98.2] | 100.0 [83.9 to 100.0] | 23.5 [6.8 to 49.9] | 95.7 [78.1 to 99.9] | 0.0 [0.0 to 24.7] | 96.8 [92.8 to 99.0] | 34.0 [21.5 to 48.3]
  Day 28, TDV-3: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-3 | 95.8 [78.9 to 99.9] | 84.6 [54.6 to 98.1] | 90.9 [70.8 to 98.9] | 92.9 [66.1 to 99.8] | 100.0 [83.9 to 100.0] | 17.6 [3.8 to 43.4] | 91.3 [72.0 to 98.9] | 0.0 [0.0 to 24.7] | 95.6 [91.1 to 98.2] | 39.6 [26.5 to 54.0]
  Day 28, TDV-4: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-4 | 79.2 [57.8 to 92.9] | 76.9 [46.2 to 95.0] | 59.1 [36.4 to 79.2] | 78.6 [49.2 to 95.3] | 85.7 [63.7 to 97.0] | 11.8 [1.5 to 36.4] | 69.6 [47.1 to 86.8] | 0.0 [0.0 to 24.7] | 74.1 [66.5 to 80.7] | 35.8 [23.1 to 50.2]
  Day 90, TDV-1: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-1 | 100.0 [85.2 to 100.0] | 92.3 [64.0 to 99.8] | 90.9 [70.8 to 98.9] | 85.7 [57.2 to 98.2] | 95.2 [76.2 to 99.9] | 17.6 [3.8 to 43.4] | 95.5 [77.2 to 99.9] | 0.0 [0.0 to 28.5] | 99.4 [96.5 to 100.0] | 41.5 [28.1 to 55.9]
  Day 90, TDV-2: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-2 | 100.0 [85.2 to 100.0] | 84.6 [54.6 to 98.1] | 90.9 [70.8 to 98.9] | 85.7 [57.2 to 98.2] | 100.0 [83.9 to 100.0] | 17.6 [3.8 to 43.4] | 100.0 [84.6 to 100.0] | 0.0 [0.0 to 28.5] | 98.7 [95.5 to 99.8] | 34.0 [21.5 to 48.3]
  Day 90, TDV-3: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 21 | 11 | 159 | 53
  Day 90, TDV-3 | 95.7 [78.1 to 99.9] | 100.0 [75.3 to 100.0] | 90.9 [70.8 to 98.9] | 85.7 [57.2 to 98.2] | 100 [83.9 to 100] | 17.6 [3.8 to 43.4] | 81.8 [59.7 to 94.8] | 9.1 [0.2 to 41.3] | 89.9 [84.2 to 94.1] | 34.0 [21.5 to 48.3]
  Day 90, TDV-4: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-4 | 82.6 [61.2 to 95.0] | 69.2 [38.6 to 90.9] | 77.3 [54.6 to 92.2] | 78.6 [49.2 to 95.3] | 66.7 [43.0 to 85.4] | 11.8 [1.5 to 36.4] | 63.6 [40.7 to 82.8] | 9.1 [0.2 to 41.3] | 69.8 [62.0 to 76.8] | 35.8 [23.1 to 50.2]
  Day 180, TDV-1: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-1 | 100.0 [83.2 to 100.0] | 91.7 [61.5 to 99.8] | 95.2 [76.2 to 99.9] | 85.7 [57.2 to 98.2] | 100.0 [83.9 to 100.0] | 23.5 [6.8 to 49.9] | 100.0 [84.6 to 100.0] | 0.0 [0.0 to 28.5] |  |
  Day 180, TDV-2: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-2 | 100.0 [83.2 to 100.0] | 83.3 [51.6 to 97.9] | 95.2 [76.2 to 99.9] | 85.7 [57.2 to 98.2] | 100.0 [83.9 to 100.0] | 23.5 [6.8 to 49.9] | 100.0 [84.6 to 100.0] | 0.0 [0.0 to 28.5] |  |
  Day 180, TDV-3: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-3 | 100.0 [83.2 to 100.0] | 91.7 [61.5 to 99.8] | 95.2 [76.2 to 99.9] | 85.7 [57.2 to 98.2] | 100.0 [83.9 to 100.0] | 35.3 [14.2 to 61.7] | 95.5 [77.2 to 99.9] | 9.1 [0.2 to 41.3] |  |
  Day 180, TDV-4: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-4 | 90.0 [68.3 to 98.8] | 66.7 [34.9 to 90.1] | 76.2 [52.8 to 91.8] | 78.6 [49.2 to 95.3] | 81.0 [58.1 to 94.6] | 17.6 [3.8 to 43.4] | 77.3 [54.6 to 92.2] | 0.0 [0.0 to 28.5] |  |
  Day 360, TDV-1: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-1 | 100.0 [82.4 to 100.0] | 91.7 [61.5 to 99.8] | 90.5 [69.6 to 98.8] | 84.6 [54.6 to 98.1] | 95.2 [76.2 to 99.9] | 29.4 [10.3 to 56.0] | 100.0 [84.6 to 100.0] | 9.1 [0.2 to 41.3] |  |
  Day 360, TDV-2: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-2 | 100.0 [82.4 to 100.0] | 83.3 [51.6 to 97.9] | 95.2 [76.2 to 99.9] | 84.6 [54.6 to 98.1] | 95.2 [76.2 to 99.9] | 29.4 [10.3 to 56.0] | 100.0 [84.6 to 100.0] | 0.0 [0.0 to 28.5] |  |
  Day 360, TDV-3: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-3 | 89.5 [66.9 to 98.7] | 83.3 [51.6 to 97.9] | 81.0 [58.1 to 94.6] | 84.6 [54.6 to 98.1] | 95.2 [76.2 to 99.9] | 29.4 [10.3 to 56.0] | 95.5 [77.2 to 99.9] | 0.0 [0.0 to 28.5] |  |
  Day 360, TDV-4: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-4 | 84.2 [60.4 to 96.6] | 75.0 [42.8 to 94.5] | 66.7 [43.0 to 85.4] | 84.6 [54.6 to 98.1] | 61.9 [38.4 to 81.9] | 17.6 [3.8 to 43.4] | 63.6 [40.7 to 82.8] | 0.0 [0.0 to 28.5] |  |
  Day 720, TDV-1: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-1 | 100.0 [79.4 to 100.0] | 100.0 [66.4 to 100.0] | 89.5 [66.9 to 98.7] | 84.6 [54.6 to 98.1] | 100.0 [83.9 to 100.0] | 23.5 [6.8 to 49.9] | 100.0 [84.6 to 100.0] | 10.0 [0.3 to 44.5] |  |
  Day 720, TDV-2: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-2 | 100.0 [79.4 to 100.0] | 88.9 [51.8 to 99.7] | 94.7 [74.0 to 99.9] | 84.6 [54.6 to 98.1] | 100.0 [83.9 to 100.0] | 23.5 [6.8 to 49.9] | 100.0 [84.6 to 100.0] | 10.0 [0.3 to 44.5] |  |
  Day 720, TDV-3: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-3 | 87.5 [61.7 to 98.4] | 88.9 [51.8 to 99.7] | 68.4 [43.4 to 87.4] | 84.6 [54.6 to 98.1] | 71.4 [47.8 to 88.7] | 17.6 [3.8 to 43.4] | 90.9 [70.8 to 98.9] | 10.0 [0.3 to 44.5] |  |
  Day 720, TDV-4: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-4 | 81.3 [54.4 to 96.0] | 77.8 [40.0 to 97.2] | 63.2 [38.4 to 83.7] | 84.6 [54.6 to 98.1] | 57.1 [34.0 to 78.2] | 23.5 [6.8 to 49.9] | 72.7 [49.8 to 89.3] | 10.0 [0.3 to 44.5] |  |
  Day 1080, TDV-1: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-1 | 100.0 [78.2 to 100.0] | 100.0 [63.1 to 100.0] | 94.4 [72.7 to 99.9] | 81.8 [48.2 to 97.7] | 95.2 [76.2 to 99.9] | 23.5 [6.8 to 49.9] | 100.0 [83.9 to 100.0] | 11.1 [0.3 to 48.2] |  |
  Day 1080, TDV-2: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-2 | 100.0 [78.2 to 100.0] | 87.5 [47.3 to 99.7] | 100.0 [81.5 to 100.0] | 81.8 [48.2 to 97.7] | 100.0 [83.9 to 100.0] | 23.5 [6.8 to 49.9] | 95.2 [76.2 to 99.9] | 0.0 [0.0 to 33.6] |  |
  Day 1080, TDV-3: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-3 | 93.3 [68.1 to 99.8] | 87.5 [47.3 to 99.7] | 77.8 [52.4 to 93.6] | 81.8 [48.2 to 97.7] | 85.7 [63.7 to 97.0] | 23.5 [6.8 to 49.9] | 95.2 [76.2 to 99.9] | 11.1 [0.3 to 48.2] |  |
  Day 1080, TDV-4: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-4 | 80.0 [51.9 to 95.7] | 87.5 [47.3 to 99.7] | 61.1 [35.7 to 82.7] | 72.7 [39.0 to 94.0] | 42.9 [21.8 to 66.0] | 17.6 [3.8 to 43.4] | 47.6 [25.7 to 70.2] | 11.1 [0.3 to 48.2] |  |

11. Secondary Outcome: Seroconversion Rate to Each of the Four Dengue Serotypes
Description: Seroconversion rate was defined as the percentage of participants with microneutralization test 50% (MNT50) titer ≥10 or, if the titer on Day 0 was ≥10, a 4-fold rise in antibody titer.
Time Frame: Day 28, 90 and 120 (Parts 1 and 2) and Days 180, 360, 720 and 1080 in Part 1
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53
percentage of participants
  Day 28, TDV-1: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-1 | 45.8 [25.6 to 67.2] | 7.7 [0.2 to 36.0] | 63.6 [40.7 to 82.8] | 0.0 [0.0 to 23.2] | 90.5 [69.6 to 98.8] | 5.9 [0.1 to 28.7] | 87.0 [66.4 to 97.2] | 7.7 [0.2 to 36.0] | 86.1 [79.7 to 91.1] | 1.9 [0.0 to 10.1]
  Day 28, TDV-2: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-2 | 33.3 [15.6 to 55.3] | 15.4 [1.9 to 45.4] | 59.1 [36.4 to 79.3] | 0.0 [0.0 to 23.2] | 85.7 [63.7 to 97.0] | 11.8 [1.5 to 36.4] | 87.0 [66.4 to 97.2] | 0.0 [0.0 to 24.7] | 86.7 [80.4 to 91.6] | 0.0 [0.0 to 6.7]
  Day 28, TDV-3: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-3 | 33.3 [15.6 to 55.3] | 0.0 [0.0 to 24.7] | 63.6 [40.7 to 82.8] | 7.1 [0.2 to 33.9] | 90.5 [69.6 to 98.8] | 0.0 [0.0 to 19.5] | 78.3 [56.3 to 92.5] | 0.0 [0.0 to 24.7] | 82.3 [75.4 to 87.9] | 1.9 [0.0 to 10.1]
  Day 28, TDV-4: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-4 | 20.8 [7.1 to 42.2] | 15.4 [1.9 to 45.4] | 31.8 [13.9 to 54.9] | 0.0 [0.0 to 23.2] | 71.4 [47.8 to 88.7] | 5.9 [0.1 to 28.7] | 60.9 [38.5 to 80.3] | 0.0 [0.0 to 24.7] | 62.7 [54.6 to 70.2] | 5.7 [1.2 to 15.7]
  Day 90, TDV-1: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-1 | 39.1 [19.7 to 61.5] | 15.4 [1.9 to 45.4] | 54.5 [32.2 to 75.6] | 7.1 [0.2 to 33.9] | 81.0 [58.1 to 94.6] | 0.0 [0.0 to 19.5] | 81.8 [59.7 to 94.8] | 0.0 [0.0 to 28.5] | 82.4 [75.6 to 88.0] | 3.8 [0.5 to 13.0]
  Day 90, TDV-2: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-2 | 30.4 [13.2 to 52.9] | 15.4 [1.9 to 45.4] | 59.1 [36.4 to 79.3] | 7.1 [0.2 to 33.9] | 85.7 [63.7 to 97.0] | 0.0 [0.0 to 19.5] | 90.9 [70.8 to 98.9] | 0.0 [0.0 to 28.5] | 86.2 [79.8 to 91.1] | 1.9 [0.0 to 10.1]
  Day 90, TDV-3: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-3 | 30.4 [13.2 to 52.9] | 23.1 [5.0 to 53.8] | 59.1 [36.4 to 79.3] | 14.3 [1.8 to 42.8] | 81.0 [58.1 to 94.6] | 0.0 [0.0 to 19.5] | 63.6 [40.7 to 82.8] | 9.1 [0.2 to 41.3] | 76.1 [68.7 to 82.5] | 0.0 [0.0 to 6.7]
  Day 90, TDV-4: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-4 | 21.7 [7.5 to 43.7] | 0.0 [0.0 to 24.7] | 50.0 [28.2 to 71.8] | 21.4 [4.7 to 50.8] | 61.9 [38.4 to 81.9] | 5.9 [0.1 to 28.7] | 54.5 [32.2 to 75.6] | 9.1 [0.2 to 41.3] | 57.9 [49.8 to 65.6] | 5.7 [1.2 to 15.7]
  Day 120, TDV-1: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-1 | 45.5 [24.4 to 67.8] | 0.0 [0.0 to 24.7] | 68.2 [45.1 to 86.1] | 14.3 [1.8 to 42.8] | 90.5 [69.6 to 98.8] | 5.9 [0.1 to 28.7] | 95.5 [77.2 to 99.9] | 0.0 [0.0 to 28.5] | 88.5 [82.4 to 93.0] | 3.8 [0.5 to 13.0]
  Day 120, TDV-2: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-2 | 45.5 [24.4 to 67.8] | 0.0 [0.0 to 24.7] | 63.6 [40.7 to 82.8] | 0.0 [0.0 to 23.2] | 95.2 [76.2 to 99.9] | 5.9 [0.1 to 28.7] | 95.5 [77.2 to 99.9] | 0.0 [0.0 to 28.5] | 90.4 [84.6 to 94.5] | 3.8 [0.5 to 13.0]
  Day 120, TDV-3: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-3 | 45.5 [24.4 to 67.8] | 30.8 [9.1 to 61.4] | 68.2 [45.1 to 86.1] | 14.3 [1.8 to 42.8] | 90.5 [69.6 to 98.8] | 17.6 [3.8 to 43.4] | 95.5 [77.2 to 99.9] | 0.0 [0.0 to 28.5] | 86.5 [80.2 to 91.5] | 1.9 [0.0 to 10.1]
  Day 120, TDV-4: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-4 | 40.9 [20.7 to 63.6] | 7.7 [0.2 to 36.0] | 45.5 [24.4 to 67.8] | 14.3 [1.8 to 42.8] | 85.7 [63.7 to 97.0] | 23.5 [6.8 to 49.9] | 95.5 [77.2 to 99.9] | 0.0 [0.0 to 28.5] | 84.0 [77.3 to 89.4] | 3.8 [0.5 to 13.0]
  Day 180, TDV-1: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-1 | 50.0 [27.2 to 72.8] | 8.3 [0.2 to 38.5] | 61.9 [38.4 to 81.9] | 0.0 [0.0 to 23.2] | 95.2 [76.2 to 99.9] | 5.9 [0.1 to 28.7] | 90.9 [70.8 to 99.9] | 0.0 [0.0 to 28.5] |  |
  Day 180, TDV-2: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-2 | 60.0 [36.1 to 80.9] | 8.3 [0.2 to 38.5] | 61.9 [38.4 to 81.9] | 7.1 [0.2 to 33.9] | 95.2 [76.2 to 99.9] | 5.9 [0.1 to 28.7] | 95.5 [77.2 to 99.9] | 0.0 [0.0 to 28.5] |  |
  Day 180, TDV-3: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-3 | 40.0 [19.1 to 63.9] | 8.3 [0.2 to 38.5] | 61.9 [38.4 to 81.9] | 7.1 [0.2 to 33.9] | 90.5 [69.5 to 98.8] | 17.6 [3.8 to 43.4] | 86.4 [65.1 to 97.1] | 9.1 [0.2 to 41.3] |  |
  Day 180, TDV-4: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-4 | 45.0 [23.1 to 68.5] | 8.3 [0.2 to 38.5] | 47.6 [25.7 to 70.2] | 7.1 [0.2 to 33.9] | 81.0 [58.1 to 94.6] | 11.8 [1.5 to 36.4] | 72.7 [49.8 to 98.3] | 0.0 [0.0 to 28.5] |  |
  Day 360, TDV-1: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-1 | 52.6 [28.9 to 75.6] | 0.0 [0.0 to 26.5] | 57.1 [34.0 to 78.2] | 15.4 [1.9 to 45.4] | 85.7 [63.7 to 97.0] | 11.8 [1.5 to 36.4] | 90.9 [70.8 to 98.9] | 9.1 [0.2 to 41.3] |  |
  Day 360, TDV-2: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-2 | 47.4 [24.4 to 71.1] | 0.0 [0.0 to 26.5] | 61.9 [38.4 to 81.9] | 15.4 [1.9 to 45.4] | 76.2 [52.8 to 91.8] | 17.6 [3.8 to 43.4] | 95.5 [77.2 to 99.9] | 0.0 [0.0 to 28.5] |  |
  Day 360, TDV-3: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-3 | 36.8 [16.3 to 61.6] | 0.0 [0.0 to 26.5] | 57.1 [34.0 to 78.2] | 15.4 [1.9 to 45.4] | 76.2 [52.8 to 91.8] | 11.8 [1.5 to 36.4] | 81.8 [59.7 to 94.8] | 0.0 [0.0 to 28.5] |  |
  Day 360, TDV-4: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-4 | 42.1 [20.3 to 66.5] | 0.0 [0.0 to 26.5] | 38.1 [18.1 to 61.6] | 7.7 [0.2 to 36.0] | 57.1 [34.0 to 78.2] | 11.8 [1.5 to 36.4] | 59.1 [36.4 to 79.3] | 0.0 [0.0 to 28.5] |  |
  Day 720, TDV-1: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-1 | 50.0 [24.7 to 75.3] | 0.0 [0.0 to 33.6] | 47.4 [24.4 to 71.1] | 15.4 [1.9 to 45.4] | 95.2 [76.2 to 99.9] | 5.9 [0.1 to 28.7] | 86.4 [65.1 to 97.1] | 10.0 [0.3 to 44.5] |  |
  Day 720, TDV-2: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-2 | 50.0 [24.7 to 75.3] | 0.0 [0.0 to 33.6] | 57.9 [33.5 to 79.7] | 7.7 [0.2 to 36.0] | 85.7 [63.7 to 97.0] | 5.9 [0.1 to 28.7] | 95.5 [77.2 to 99.9] | 10.0 [0.3 to 44.5] |  |
  Day 720, TDV-3: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-3 | 43.8 [19.8 to 70.1] | 0.0 [0.0 to 33.6] | 31.6 [12.6 to 56.6] | 15.4 [1.9 to 45.4] | 66.7 [43.0 to 85.4] | 5.9 [0.1 to 28.7] | 86.4 [65.1 to 97.1] | 10.0 [0.3 to 44.5] |  |
  Day 720, TDV-4: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-4 | 18.8 [4.0 to 45.6] | 0.0 [0.0 to 36.9] | 36.8 [16.3 to 61.6] | 15.4 [1.9 to 45.4] | 47.6 [25.7 to 70.2] | 17.6 [3.8 to 43.4] | 63.6 [40.7 to 82.8] | 10.0 [0.3 to 44.5] |  |
  Day 1080, TDV-1: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-1 | 46.7 [21.3 to 73.4] | 0.0 [0.0 to 36.9] | 55.6 [30.8 to 78.5] | 18.2 [2.3 to 51.8] | 90.5 [69.6 to 98.8] | 5.9 [0.1 to 28.7] | 85.7 [63.7 to 97.0] | 11.1 [0.3 to 48.2] |  |
  Day 1080, TDV-2: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-2 | 46.7 [21.3 to 73.4] | 0.0 [0.0 to 36.9] | 61.1 [35.7 to 82.7] | 9.1 [0.2 to 41.3] | 81.0 [58.1 to 94.6] | 5.9 [0.1 to 28.7] | 85.7 [63.7 to 97.0] | 0.0 [0.0 to 33.6] |  |
  Day 1080, TDV-3: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-3 | 33.3 [11.8 to 61.6] | 0.0 [0.0 to 36.9] | 44.4 [21.5 to 69.2] | 18.2 [2.3 to 51.8] | 81.0 [58.1 to 94.6] | 5.9 [0.1 to 28.7] | 90.5 [69.6 to 98.8] | 11.1 [0.3 to 48.2] |  |
  Day 1080, TDV-4: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-4 | 13.3 [1.7 to 40.5] | 12.5 [0.3 to 52.7] | 27.8 [9.7 to 53.5] | 18.2 [2.3 to 51.8] | 33.3 [14.6 to 57.0] | 11.8 [1.5 to 36.4] | 38.1 [18.1 to 61.6] | 11.1 [0.3 to 48.2] |  |

12. Secondary Outcome: Geometric Mean Neutralizing Antibody Titers (GMTs) of All Four Dengue Serotypes
Description: GMTs were assessed for the four dengue serotypes: TDV-1, TDV-2, TDV-3, and TDV-4.
Time Frame: Day 28, 90 and 120 (Parts 1 and 2) and Days 180, 360, 720 and 1080 in Part 1
Population: The FAS included all randomized participants who received at least one dose of study vaccine and for whom valid pre-dosing and at least one valid post-dosing blood sample have been received. Here "n" is the number of participants with microneutralizing (MN) assay samples.
Measure: Mean (95% Confidence Interval); unit: titer
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53
titer
  Day 28, TDV-1: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-1 | 1156.9 [582.0 to 2299.9] | 396.1 [120.6 to 1301.2] | 919.5 [273.1 to 3096.1] | 204.9 [59.8 to 702.6] | 383.7 [178.1 to 826.5] | 11.3 [4.4 to 29.3] | 395.2 [190.0 to 822.0] | 5.3 [4.7 to 5.9] | 522.2 [396.5 to 687.7] | 28.7 [14.8 to 55.5]
  Day 28, TDV-2: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-2 | 2313.9 [1328.1 to 4031.2] | 178.0 [44.4 to 712.9] | 1726.6 [539.2 to 5528.8] | 420.2 [116.5 to 1515.6] | 2357.2 [1218.6 to 4559.7] | 13.9 [5.0 to 38.6] | 1134.6 [479.9 to 2682.6] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the lower limit of detection (LLOD). | 1496.5 [1129.1 to 1983.4] | 16.4 [9.7 to 27.9]
  Day 28, TDV-3: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-3 | 538.2 [218.3 to 1326.5] | 226.3 [70.1 to 730.7] | 330.2 [94.4 to 1155.9] | 304.5 [83.9 to 1105.6] | 314.8 [135.3 to 732.3] | 8.5 [4.1 to 17.4] | 129.6 [52.9 to 317.6] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 206.9 [149.9 to 285.7] | 19.4 [11.5 to 32.6]
  Day 28, TDV-4: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-4 | 130.7 [54.3 to 314.5] | 55.1 [15.6 to 194.9] | 56.6 [19.1 to 167.3] | 46.4 [17.6 to 122.4] | 61.4 [27.1 to 139.4] | 7.2 [3.9 to 13.4] | 27.0 [12.5 to 58.5] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 45.4 [33.2 to 62.0] | 11.0 [7.8 to 15.6]
  Day 90, TDV-1: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-1 | 961.3 [413.5 to 2235.2] | 751.0 [227.1 to 2483.1] | 555.4 [156.9 to 1966.2] | 215.3 [55.4 to 836.4] | 245.7 [82.2 to 734.7] | 10.8 [4.2 to 28.3] | 165.1 [69.4 to 392.8] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 324.2 [239.1 to 439.6] | 27.9 [14.6 to 53.4]
  Day 90, TDV-2: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-2 | 2073.1 [1267.0 to 3392.1] | 320.0 [74.2 to 1379.3] | 1146.4 [416.7 to 3153.6] | 463.9 [120.1 to 1792.0] | 966.9 [451.8 to 2069.2] | 10.0 [4.3 to 23.1] | 467.0 [205.7 to 1060.3] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 463.5 [364.0 to 590.2] | 15.2 [8.9 to 25.9]
  Day 90, TDV-3: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-3 | 510.5 [218.3 to 1194.1] | 272.7 [86.4 to 860.4] | 193.3 [54.9 to 680.7] | 336.2 [95.3 to 1185.8] | 195.0 [73.3 to 518.8] | 8.5 [4.4 to 16.5] | 66.2 [28.3 to 154.8] | 5.3 [4.6 to 6.1] | 139.5 [99.7 to 195.1] | 17.1 [10.2 to 28.5]
  Day 90, TDV-4: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-4 | 125.7 [57.7 to 274.1] | 36.0 [13.3 to 97.2] | 76.3 [29.3 to 198.9] | 69.0 [23.7 to 200.4] | 31.2 [12.3 to 79.3] | 7.5 [4.0 to 14.3] | 16.8 [9.3 to 30.5] | 5.3 [4.6 to 6.1] | 33.7 [25.4 to 44.7] | 11.8 [8.2 to 16.9]
  Day 120, TDV-1: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-1 | 1240.3 [585.2 to 2628.8] | 356.0 [117.8 to 1076.1] | 1300.3 [528.5 to 3199.4] | 164.0 [52.8 to 509.4] | 551.7 [231.6 to 1313.8] | 13.9 [4.9 to 39.2] | 582.3 [275.9 to 1229.1] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 710.4 [547.5 to 921.9] | 29.6 [15.6 to 56.1]
  Day 120, TDV-2: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-2 | 2403.7 [1443.5 to 4002.6] | 272.7 [60.9 to 1221.6] | 1754.0 [744.2 to 4134.4] | 399.9 [109.7 to 1457.7] | 983.0 [423.5 to 2281.6] | 17.3 [4.6 to 65.9] | 459.7 [232.6 to 908.7] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 605.4 [490.6 to 747.1] | 16.2 [9.5 to 27.8]
  Day 120, TDV-3: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-3 | 650.2 [288.1 to 1467.0] | 287.6 [116.7 to 709.1] | 340.8 [121.3 to 957.6] | 289.8 [82.7 to 1016.1] | 377.4 [170.3 to 836.6] | 14.4 [5.0 to 41.8] | 196.4 [115.2 to 334.8] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 332.3 [263.1 to 419.7] | 19.0 [11.3 to 32.0]
  Day 120, TDV-4: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-4 | 193.3 [84.7 to 441.1] | 36.0 [10.5 to 123.2] | 82.6 [31.8 to 214.1] | 69.0 [23.5 to 202.7] | 64.6 [27.6 to 151.1] | 13.9 [5.4 to 35.3] | 41.3 [24.9 to 68.3] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 76.5 [60.5 to 96.8] | 11.2 [8.0 to 15.9]
  Day 180, TDV-1: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-1 | 831.7 [332.7 to 2078.8] | 320.0 [86.0 to 1191.4] | 954.7 [280.8 to 3245.7] | 141.6 [38.8 to 516.4] | 230.5 [107.2 to 495.4] | 12.8 [4.7 to 34.4] | 249.2 [113.5 to 546.8] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 180, TDV-2: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-2 | 2521.2 [1444.5 to 4400.4] | 226.3 [48.9 to 1046.4] | 1515.6 [593.7 to 3869.0] | 412.3 [104.9 to 1620.6] | 642.5 [325.9 to 1266.8] | 14.4 [4.9 to 42.4] | 399.3 [194.7 to 819.1] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 180, TDV-3: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-3 | 422.2 [179.1 to 995.5] | 285.1 [74.7 to 1087.6] | 321.2 [101.3 to 1018.4] | 206.1 [65.9 to 645.0] | 189.1 [84.2 to 424.6] | 12.5 [5.5 to 28.4] | 93.6 [41.4 to 211.7] | 6.0 [4.0 to 9.2] |  |
  Day 180, TDV-4: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-4 | 146.7 [62.8 to 342.7] | 44.9 [13.0 to 155.7] | 71.5 [27.6 to 185.0] | 51.2 [19.8 to 132.4] | 47.2 [20.4 to 109.3] | 9.2 [4.4 to 19.4] | 28.3 [14.3 to 56.0] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 360, TDV-1: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-1 | 1417.4 [474.5 to 4233.5] | 320.0 [78.5 to 1304.5] | 642.5 [179.5 to 2299.8] | 221.0 [48.9 to 999.6] | 132.0 [51.6 to 338.0] | 15.7 [5.5 to 45.2] | 220.9 [90.3 to 540.2] | 5.3 [4.6 to 6.1] |  |
  Day 360, TDV-2: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-2 | 2410.7 [1120.9 to 5185.0] | 271.8 [60.9 to 1212.7] | 852.2 [369.9 to 1963.3] | 523.6 [113.4 to 2416.7] | 329.5 [161.7 to 671.1] | 17.1 [6.0 to 48.7] | 298.8 [141.1 to 632.8] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 360, TDV-3: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-3 | 537.9 [158.5 to 1825.3] | 256.2 [70.2 to 935.3] | 171.3 [51.1 to 574.0] | 209.5 [55.4 to 792.9] | 103.1 [40.0 to 265.6] | 11.8 [5.3 to 26.0] | 89.9 [43.9 to 184.1] | 5 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 360, TDV-4: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-4 | 163.6 [56.2 to 476.4] | 44.9 [13.5 to 149.1] | 73.8 [26.9 to 202.8] | 59.9 [19.4 to 184.4] | 27.0 [11.9 to 61.0] | 7.5 [4.0 to 14.0] | 20.0 [10.8 to 37.0] | 5 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 720, TDV-1: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-1 | 924.9 [289.1 to 2959.4] | 691.2 [175.7 to 2720.1] | 452.5 [124.5 to 1644.5] | 258.5 [67.0 to 997.9] | 115.0 [45.4 to 291.1] | 12.8 [4.8 to 34.2] | 248.7 [103.4 to 597.9] | 5.7 [4.2 to 7.9] |  |
  Day 720, TDV-2: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-2 | 1399.4 [704.8 to 2778.8] | 244.9 [50.1 to 1197.1] | 714.0 [247.9 to 2056.8] | 396.1 [98.3 to 1595.4] | 280.4 [135.1 to 582.2] | 13.0 [5.0 to 33.9] | 219.3 [106.7 to 450.7] | 5.4 [4.6 to 6.3] |  |
  Day 720, TDV-3: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-3 | 515.4 [140.6 to 1888.5] | 403.2 [96.0 to 1692.5] | 154.3 [36.7 to 649.1] | 303.4 [70.9 to 1297.4] | 65.6 [21.2 to 203.0] | 8.8 [4.5 to 17.5] | 104.6 [37.7 to 289.8] | 8.1 [2.7 to 24.3] |  |
  Day 720, TDV-4: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-4 | 106.0 [40.5 to 277.3] | 48.5 [13.1 to 180.2] | 66.7 [22.5 to 197.2] | 93.9 [29.0 to 303.8] | 24.4 [10.8 to 55.2] | 8.5 [4.7 to 15.2] | 26.6 [12.3 to 57.3] | 5.7 [4.2 to 7.9] |  |
  Day 1080, TDV-1: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-1 | 718.4 [239.3 to 2156.7] | 905.1 [243.2 to 3368.4] | 508.0 [137.6 to 1874.9] | 219.3 [41.2 to 1165.6] | 92.8 [36.5 to 236.2] | 12.8 [4.8 to 34.2] | 149.8 [63.9 to 351.1] | 6.3 [3.7 to 10.7] |  |
  Day 1080, TDV-2: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-2 | 702.0 [403.1 to 1222.4] | 146.7 [27.3 to 787.7] | 615.8 [277.5 to 1366.8] | 256.7 [61.0 to 1079.3] | 160.0 [76.5 to 334.8] | 12.8 [5.2 to 31.7] | 118.9 [57.0 to 248.0] | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 1080, TDV-3: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-3 | 291.8 [82.5 to 1032.3] | 472.6 [84.6 to 2641.0] | 201.6 [54.6 to 744.0] | 264.9 [53.4 to 1313.1] | 70.1 [27.6 to 178.4] | 9.6 [4.6 to 20.1] | 80.0 [31.9 to 200.7] | 9.3 [2.2 to 38.3] |  |
  Day 1080, TDV-4: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-4 | 81.9 [30.9 to 216.9] | 80.0 [17.5 to 364.8] | 61.1 [21.7 to 172.3] | 80.0 [18.9 to 338.6] | 17.5 [8.4 to 36.6] | 7.2 [4.2 to 12.3] | 17.0 [8.6 to 33.3] | 5.4 [4.5 to 6.4] |  |

13. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Dengue Neutralizing Antibody Titers for Each of the 4 Dengue Serotypes
Time Frame: Day 28 and Day 90 (Parts 1 and 2) and Days 120, 180, 360, 720 and 1080 in Part 1
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53
fold rise
  Day 28, TDV-1: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-1 | 3.41 [1.61 to 7.24] | 0.90 [0.57 to 1.41] | 8.93 [3.61 to 22.09] | 1.03 [0.67 to 1.56] | 29.47 [11.70 to 74.22] | 1.00 [0.88 to 1.13] | 27.94 [13.64 to 57.23] | 1.05 [0.94 to 1.18] | 27.58 [20.91 to 36.38] | 0.97 [0.82 to 1.16]
  Day 28, TDV-2: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-2 | 7.89 [2.01 to 31.00] | 0.71 [0.45 to 1.11] | 20.26 [5.34 to 76.93] | 1.05 [0.69 to 1.59] | 181.02 [47.86 to 684.60] | 1.39 [0.81 to 2.37] | 128.00 [44.62 to 367.22] | 1.00 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the lower limit of detection (LLOD). | 113.02 [0.1 to 8192.0] | 0.94 [0.0 to 2.0]
  Day 28, TDV-3: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-3 | 2.34 [1.22 to 4.52] | 0.97 [0.74 to 1.28] | 4.40 [1.85 to 10.48] | 1.08 [0.71 to 1.63] | 24.17 [10.16 to 57.49] | 1.02 [0.98 to 1.07] | 13.76 [6.01 to 31.50] | 1.00 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 12.47 [9.18 to 16.92] | 0.82 [0.71 to 0.94]
  Day 28, TDV-4: number analyzed (Participants) | 24 | 13 | 22 | 14 | 21 | 17 | 23 | 13 | 158 | 53
  Day 28, TDV-4 | 1.71 [0.88 to 3.31] | 1.11 [0.65 to 1.90] | 2.74 [1.11 to 6.80] | 0.82 [0.53 to 1.26] | 7.49 [3.60 to 15.58] | 1.13 [0.94 to 1.36] | 4.00 [1.85 to 8.66] | 0.95 [0.84 to 1.06] | 74.1 [66.5 to 80.7] | 35.8 [23.1 to 50.2]
  Day 90, TDV-1: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-1 | 3.10 [1.26 to 7.59] | 1.70 [0.75 to 3.90] | 5.40 [2.50 to 11.63] | 1.08 [0.71 to 1.63] | 18.87 [7.61 to 46.81] | 0.96 [0.88 to 1.05] | 11.14 [5.37 to 23.09] | 1.000 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 324.2 [239.1 to 439.6] | 27.9 [14.6 to 53.4]
  Day 90, TDV-2: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-2 | 7.09 [2.20 to 22.83] | 1.27 [0.78 to 2.08] | 13.45 [4.52 to 40.08] | 1.16 [0.74 to 1.83] | 74.25 [30.35 to 181.64] | 1.00 [0.88 to 1.13] | 51.33 [20.33 to 129.62] | 1.00 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 463.5 [364.0 to 590.2] | 15.2 [8.9 to 25.9]
  Day 90, TDV-3: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-3 | 2.29 [1.29 to 4.05] | 1.17 [0.74 to 1.85] | 2.57 [1.14 to 5.80] | 1.19 [0.67 to 2.13] | 14.98 [6.11 to 36.75] | 1.02 [0.92 to 1.13] | 6.83 [3.13 to 14.93] | 1.07 [0.93 to 1.23] | 139.5 [99.7 to 195.1] | 17.1 [10.2 to 28.5]
  Day 90, TDV-4: number analyzed (Participants) | 23 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 159 | 53
  Day 90, TDV-4 | 1.64 [1.02 to 2.66] | 0.73 [0.52 to 1.01] | 3.70 [1.78 to 7.66] | 1.22 [0.72 to 2.07] | 3.81 [1.73 to 8.36] | 1.18 [0.90 to 1.54] | 2.45 [1.39 to 4.32] | 1.00 [0.81 to 1.23] | 33.7 [25.4 to 44.7] | 11.8 [8.2 to 16.9]
  Day 120, TDV-1: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-1 | 3.64 [1.09 to 12.10] | 0.81 [0.56 to 1.16] | 12.63 [5.56 to 28.70] | 0.82 [0.34 to 2.01] | 42.36 [19.57 to 91.70] | 1.23 [0.72 to 2.09] | 39.27 [24.12 to 63.94] | 1.00 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 35.44 [26.46 to 47.48] | 1.01 [0.79 to 1.28]
  Day 120, TDV-2: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-2 | 8.79 [2.81 to 27.47] | 1.08 [0.79 to 1.49] | 20.59 [6.45 to 65.66] | 1.00 [0.67 to 1.50] | 75.48 [29.82 to 191.08] | 1.73 [0.56 to 5.38] | 50.53 [24.11 to 105.89] | 1.00 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 44.16 [33.51 to 58.20] | 0.92 [0.67 to 1.28]
  Day 120, TDV-3: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-3 | 2.78 [1.44 to 5.37] | 1.24 [0.70 to 2.20] | 4.54 [2.02 to 10.17] | 1.03 [0.60 to 1.75] | 28.98 [14.52 to 57.87] | 1.73 [0.73 to 4.14] | 20.26 [12.02 to 34.17] | 1.00 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 19.20 [14.75 to 24.98] | 0.80 [0.64 to 1.01]
  Day 120, TDV-4: number analyzed (Participants) | 22 | 13 | 22 | 14 | 21 | 17 | 22 | 11 | 156 | 53
  Day 120, TDV-4 | 2.45 [1.44 to 4.19] | 0.73 [0.43 to 1.23] | 4.00 [2.00 to 8.00] | 1.22 [0.72 to 2.07] | 7.87 [4.25 to 14.57] | 2.17 [0.99 to 4.76] | 6.02 [3.81 to 9.53] | 0.94 [0.82 to 1.08] | 7.43 [5.96 to 9.27] | 1.03 [0.91 to 1.16]
  Day 180, TDV-1: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-1 | 3.94 [1.35 to 11.54] | 0.89 [0.59 to 1.35] | 9.16 [2.89 to 29.05] | 0.71 [0.45 to 1.10] | 17.70 [10.04 to 31.22] | 1.13 [0.77 to 1.66] | 16.81 [9.56 to 29.53] | 1.00 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 180, TDV-2: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-2 | 11.53 [3.61 to 36.83] | 0.94 [0.55 to 1.63] | 17.16 [5.15 to 57.17] | 1.03 [0.58 to 1.84] | 49.34 [22.02 to 110.57] | 1.44 [0.66 to 3.17] | 43.89 [21.22 to 90.80] | 1.00 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 180, TDV-3: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-3 | 2.42 [1.23 to 4.76] | 1.26 [0.95 to 1.68] | 4.58 [1.72 to 12.21] | 0.73 [0.44 to 1.20] | 14.52 [7.70 to 27.38] | 1.50 [0.86 to 2.64] | 9.66 [4.84 to 19.30] | 1.21 [0.79 to 1.84] |  |
  Day 180, TDV-4: number analyzed (Participants) | 20 | 12 | 21 | 14 | 21 | 17 | 22 | 11 | 0 | 0
  Day 180, TDV-4 | 2.38 [1.43 to 3.95] | 1.00 [0.63 to 1.58] | 3.35 [1.60 to 7.01] | 0.91 [0.60 to 1.37] | 5.76 [3.14 to 10.55] | 1.44 [0.88 to 2.36] | 4.13 [2.29 to 7.43] | 0.94 [0.82 to 1.08] |  |
  Day 360, TDV-1: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-1 | 5.51 [2.13 to 14.26] | 0.67 [0.47 to 0.95] | 6.17 [2.36 to 16.14] | 1.09 [0.50 to 2.37] | 10.14 [4.81 to 21.39] | 1.39 [0.91 to 2.12] | 14.90 [7.48 to 29.66] | 1.07 [0.93 to 1.23] |  |
  Day 360, TDV-2: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-2 | 9.04 [2.76 to 29.60] | 0.93 [0.64 to 1.34] | 9.65 [3.34 to 27.83] | 1.16 [0.54 to 2.46] | 25.30 [10.10 to 63.38] | 1.71 [0.81 to 3.59] | 32.84 [15.76 to 68.42] | 1.00 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 360, TDV-3: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-3 | 2.56 [1.21 to 5.39] | 0.95 [0.71 to 1.27] | 2.44 [1.00 to 5.96] | 0.83 [0.44 to 1.57] | 7.92 [3.28 to 19.10] | 1.41 [0.88 to 2.29] | 9.28 [4.55 to 18.92] | 1.00 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 360, TDV-4: number analyzed (Participants) | 19 | 12 | 21 | 13 | 21 | 17 | 22 | 11 | 0 | 0
  Day 360, TDV-4 | 2.32 [1.15 to 4.70] | 0.75 [0.53 to 1.06] | 3.45 [1.66 to 7.17] | 1.03 [0.45 to 2.38] | 3.29 [1.83 to 5.89] | 1.18 [0.96 to 1.44] | 2.92 [1.71 to 4.98] | 0.94 [0.82 to 1.08] |  |
  Day 720, TDV-1: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-1 | 4.65 [1.45 to 14.97] | 0.63 [0.43 to 0.92] | 3.65 [1.68 to 7.96] | 1.27 [0.64 to 2.54] | 8.83 [4.69 to 16.64] | 1.13 [0.87 to 1.46] | 16.77 [7.12 to 39.51] | 1.15 [0.84 to 1.57] |  |
  Day 720, TDV-2: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-2 | 9.13 [2.52 to 33.07] | 0.80 [0.51 to 1.24] | 8.61 [3.28 to 22.56] | 0.88 [0.52 to 1.48] | 21.53 [9.91 to 46.81] | 1.30 [0.73 to 2.32] | 24.10 [11.73 to 49.52] | 1.07 [0.92 to 1.25] |  |
  Day 720, TDV-3: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-3 | 3.15 [1.38 to 7.21] | 0.93 [0.67 to 1.28] | 2.00 [0.76 to 5.28] | 1.21 [0.72 to 2.02] | 5.04 [2.21 to 11.50] | 1.06 [0.80 to 1.41] | 10.79 [4.16 to 28.00] | 1.62 [0.54 to 4.87] |  |
  Day 720, TDV-4: number analyzed (Participants) | 16 | 9 | 19 | 13 | 21 | 17 | 22 | 10 | 0 | 0
  Day 720, TDV-4 | 1.54 [0.77 to 3.10] | 0.56 [0.39 to 0.82] | 2.88 [1.41 to 5.90] | 1.62 [0.76 to 3.43] | 2.97 [1.56 to 5.66] | 1.33 [0.95 to 1.86] | 3.88 [1.89 to 7.96] | 1.07 [0.74 to 1.55] |  |
  Day 1080, TDV-1: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-1 | 3.91 [1.40 to 10.94] | 0.77 [0.45 to 1.31] | 3.43 [1.66 to 7.08] | 1.33 [0.73 to 2.41] | 7.13 [3.86 to 13.17] | 1.13 [0.79 to 1.62] | 9.59 [4.72 to 19.48] | 1.26 [0.74 to 2.15] |  |
  Day 1080, TDV-2: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-2 | 4.59 [1.45 to 14.59] | 0.68 [0.51 to 0.90] | 6.35 [2.54 to 15.87] | 0.83 [0.51 to 1.34] | 12.29 [5.76 to 26.22] | 1.28 [0.73 to 2.24] | 12.70 [5.92 to 27.25] | 1.00 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. |  |
  Day 1080, TDV-3: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-3 | 1.87 [0.98 to 3.54] | 1.04 [0.75 to 1.45] | 2.33 [0.97 to 5.59] | 1.17 [0.65 to 2.10] | 5.38 [2.71 to 10.71] | 1.15 [0.89 to 1.50] | 8.55 [3.97 to 18.38] | 1.85 [0.45 to 7.67] |  |
  Day 1080, TDV-4: number analyzed (Participants) | 15 | 8 | 18 | 11 | 21 | 17 | 21 | 9 | 0 | 0
  Day 1080, TDV-4 | 1.15 [0.71 to 1.87] | 1.00 [0.58 to 1.71] | 2.42 [1.18 to 4.98] | 1.46 [0.66 to 3.21] | 2.14 [1.23 to 3.72] | 1.13 [0.94 to 1.36] | 2.44 [1.40 to 4.25] | 1.00 [0.77 to 1.31] |  |

14. Secondary Outcome: Number of Participants With Confirmed Dengue Fever
Description: Dengue fever was assessed in participants who had 3 consecutive days of fever >38°C and tested positive for dengue virus by polymerase chain reaction (PCR) analysis.
Time Frame: Day 1 to Day 1080
Population: The safety set included all randomized participants who received at least one dose of study vaccine (or placebo).
Measure: Number; unit: participants
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Number analyzed (Participants) | 24 | 14 | 22 | 14 | 21 | 17 | 23 | 13 | 159 | 53
participants | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: Serious AEs were collected throughout the study Day 0 up to Day 1080. Other (non-serious) AEs were collected within 28 days of all vaccinations (up to Day 28 and Day 118).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part I: TDV 21 to 45 Years | Part I: Placebo 21 to 45 Years | Part I: TDV 12 to 20 Years | Part I: Placebo 12 to 20 Years | Part I: TDV 6 to 11 Years | Part I: Placebo 6 to 11 Years | Part I: TDV 1.5 to 5 Years | Part I: Placebo 1.5 to 5 Years | Part II: TDV 1.5 to 11 Years | Part II: Placebo 1.5 to 11 Years
Serious Adverse Events (participants affected / at risk) | 4/24 | 0/14 | 1/22 | 0/14 | 4/21 | 1/17 | 1/23 | 2/13 | 14/159 | 2/53
Other Adverse Events (participants affected / at risk) | 11/24 | 7/14 | 13/22 | 8/14 | 9/21 | 11/17 | 14/23 | 12/13 | 87/159 | 30/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: TDV 21 to 45 Years (N=24) | Part I: Placebo 21 to 45 Years (N=14) | Part I: TDV 12 to 20 Years (N=22) | Part I: Placebo 12 to 20 Years (N=14) | Part I: TDV 6 to 11 Years (N=21) | Part I: Placebo 6 to 11 Years (N=17) | Part I: TDV 1.5 to 5 Years (N=23) | Part I: Placebo 1.5 to 5 Years (N=13) | Part II: TDV 1.5 to 11 Years (N=159) | Part II: Placebo 1.5 to 11 Years (N=53)
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Child maltreatment syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: TDV 21 to 45 Years (N=24) | Part I: Placebo 21 to 45 Years (N=14) | Part I: TDV 12 to 20 Years (N=22) | Part I: Placebo 12 to 20 Years (N=14) | Part I: TDV 6 to 11 Years (N=21) | Part I: Placebo 6 to 11 Years (N=17) | Part I: TDV 1.5 to 5 Years (N=23) | Part I: Placebo 1.5 to 5 Years (N=13) | Part II: TDV 1.5 to 11 Years (N=159) | Part II: Placebo 1.5 to 11 Years (N=53)
Headache (Nervous system disorders) | 4 | 3 | 7 | 1 | 4 | 3 | 1 | 0 | 13 | 3
Laryngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 8 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 6 | 2
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 1 | 16 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 3 | 2 | 8 | 7 | 32 | 14
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 4 | 0 | 0 | 1 | 0 | 2 | 0
Injection site pain (General disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Injection site erythema (General disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 6 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 1 | 11 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.